CLINICAL TRIAL: NCT00293956
Title: Thyroid Function in Term and Near Term Infants With Respiratory Distress and Its' Relation to Severity of Illness
Brief Title: Thyroid Function in Term Infants With Respiratory Distress
Status: Completed | Type: Observational
Sponsor: Christiana Care Health Services (Other)
Responsible Party: David A. Paul, MD, Christiana Hospital
Other Study IDs: 25190
Record Dates: First submitted 2006-02-16; First posted 2006-02-20 (Estimated); Last update posted 2008-01-18 (Estimated); Status verified 2008-01

CONDITIONS: Transient Hypothyroxinemia; Infant, Newborn
Keywords: hypothyroxinemia; full term infants; near term infants; respiratory distress; thyroid disease
MeSH Terms: conditions — Dyspnea; Thyroid Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Full-term and near-term infants with respiratory distress in the first 24 hours of life

SUMMARY:
This study was designed to evaluate the level of certain hormones (thyroid hormones and cortisol) in full term or close to full term infants who have respiratory distress severe enough to require respiratory support. The purpose of this study is to determine if there is a relationship between these hormone levels and how sick these infants are who require help with breathing following birth.

Hypothesis: Infants who are born full term or near full term and who have low hormone levels will have higher severity of illness.

DETAILED DESCRIPTION:
Transient hypothyroxinemia, as demonstrated by low T4 and free T4 levels with normal levels of TSH, in preterm infants has been associated with increased severity of illness and adverse outcomes. Effects of thyroid function in term infants is less well studied. Previous research in the Special Care Nursery at Christiana Hospital has indicated that transient hypothyroxinemia in intubated term infants was associated with increased severity of illness and the need for more intensive rescue therapies. However, free T4, the biologically active substance was not measured in our previous study.

Infants who meet criteria for the study will begin participation after parental informed consent is obtained. Infants who are enrolled will have serial measurements of thyroid stimulating hormone (TSH), T4, free T4, free T3, and cortisol. These measurements will be obtained at four specific time intervals throughout the first week of the infant's life. The medical team will be blinded to the results of the hormone testing. The results will be reviewed by an unblinded study investigator and an endocrinologist will be consulted if abnormal results are reported.

These hormone levels will be compared with severity of illness and level of respiratory support needed in order to establish an association between thyroid function and illness severity. Illness severity will be quantified by using the Score for Neonatal Acute Physiology (SNAP). SNAP scores require collecting data from vital signs and results of labs that are considered standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Infants born > or = to 35 weeks gestation
* Infants admitted to the neonatal intensive care unit at Christiana Hospital
* Respiratory distress requiring use of mechanical ventilation or nasal CPAP (continuous positive airway pressure)
* Parental informed consent

Exclusion Criteria:

* Infants born < 35 weeks gestation
* Infants with documented congenital abnormalities which directly impact the cardiorespiratory system

Max Age: 6 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Full-term and near-term infants with respiratory distress during the first 24 hours of life.
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2006-01; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
To determine if thyroid function, particularly free T4, is associated with severity of illness in term and near term infants with respiratory distress who require endotracheal intubation or nasal CPAP. | Birth until 120 hours of life

CONTACTS AND LOCATIONS:
Overall Officials: David A. Paul, MD, Principal Investigator — Christiana Care Health Systems; Erika M. Yencha, MD, Principal Investigator — Christiana Care Health Systems
Locations (1):
- Christiana Hospital, Newark, Delaware, United States

REFERENCES:
- [Background] Huang CB, Chen FS, Chung MY. Transient hypothyroxinemia of prematurity is associated with abnormal cranial ultrasound and illness severity. Am J Perinatol. 2002 Apr;19(3):139-47. doi: 10.1055/s-2002-25308. PMID 12012289
- [Background] Paul DA, Leef KH, Voss B, Stefano JL, Bartoshesky L. Thyroxine and illness severity in very low-birth-weight infants. Thyroid. 2001 Sep;11(9):871-5. doi: 10.1089/105072501316973136. PMID 11575857
- [Background] Lim DJ, Herring MK, Leef KH, Getchell J, Bartoshesky LE, Paul DA. Hypothyroxinemia in mechanically ventilated term infants is associated with increased use of rescue therapies. Pediatrics. 2005 Feb;115(2):406-10. doi: 10.1542/peds.2004-0192. PMID 15687450
- [Background] Watterberg KL, Gerdes JS, Cook KL. Impaired glucocorticoid synthesis in premature infants developing chronic lung disease. Pediatr Res. 2001 Aug;50(2):190-5. doi: 10.1203/00006450-200108000-00005. PMID 11477202
- [Background] Simpson J, Williams FL, Delahunty C, van Toor H, Wu SY, Ogston SA, Visser TJ, Hume R; Scottish Preterm Thyroid Group. Serum thyroid hormones in preterm infants and relationships to indices of severity of intercurrent illness. J Clin Endocrinol Metab. 2005 Mar;90(3):1271-9. doi: 10.1210/jc.2004-2091. Epub 2004 Dec 21. PMID 15613404
- [Background] Richardson DK, Gray JE, McCormick MC, Workman K, Goldmann DA. Score for Neonatal Acute Physiology: a physiologic severity index for neonatal intensive care. Pediatrics. 1993 Mar;91(3):617-23. PMID 8441569